CLINICAL TRIAL: NCT00514540
Title: Phase II Study of Carboplatin Plus Docetaxel (Taxotere) in Patients With Anaplastic Prostate Carcinoma
Brief Title: Carboplatin Plus Docetaxel (Taxotere) in Anaplastic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0097
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Anaplastic Prostate Cancer; Carboplatin; Docetaxel; Taxotere; Paraplatin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Carboplatin; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- First-Line/Second-Line Chemotherapy (Experimental): First-Line (CD) Chemotherapy: Carboplatin area under the curve (AUC) = 5, intravenous (IV) over 30 minutes and Docetaxel 75 mg/m^2 IV over 60 minutes, Day 1. Repeated every 3 weeks.
  Second-Line (EP) Chemotherapy: Etoposide 120 mg/m^2 daily for 3 days and Cisplatin 25 mg/m^2 for 3 days with adequate intravenous hydration mannitol diuresis and supportive care (antiemetics). Repeated every 3 weeks.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m^2 IV over 60 Minutes on Day 1 of 21 day cycle.
  Other Names: Taxotere
Drug: Carboplatin — AUC = 5 IV Over 30 Minutes On Day 1 of 21 day cycle.
  Other Names: Paraplatin
Drug: Etoposide — 120 mg/m^2 daily for 3 days of 21 day cycle.
Drug: Cisplatin — 25 mg/m^2 for 3 days of 21 day cycle.

SUMMARY:
The goal of this clinical research study is to learn about how effective 2 chemotherapy drugs carboplatin (Paraplatin) plus docetaxel (Taxotere) in the treatment of patients with anaplastic prostate cancer. Patients who continue to have advanced disease will be switched to etoposide (VePesid) plus cisplatin (Platinol-AQ) to study how effective this second line of chemotherapy is in the treatment of patients iwth anaplastic prostate cancer.

The side effects, characteristics of patients who respond, and overall survival will also be studied.

DETAILED DESCRIPTION:
Carboplatin is designed to interfere with the growth of cancer cells by stopping cell division.

Docetaxel is designed to stop the growth of cancer cells, which may cause the cells to die. It is believed to be weakly effective at killing blood vessels in cancer cells as well.

Etoposide is a drug that has been shown to interfere with the growth of cancer cells, which may cause them to eventually die.

Cisplatin has an atom at its center that contains platinum. The platinum is supposed to poison the cancer cells, which may cause them to eventually die.

If you are found to be eligible to take part in this study, you will receive carboplatin plus docetaxel by a vein or central line in a vein. You will receive carboplatin over about 30 minutes and docetaxel over about 60 minutes. You will receive this therapy combination on Day 1 of each cycle of therapy (every 3-4 weeks), depending on the recovery of your bone marrow. These 3-4 weeks are considered 1 cycle of therapy. This therapy combination will be given on an outpatient basis. If you experience any side effects, your dose of docetaxel plus carboplatin may be decreased.

You will be given dexamethasone, by a vein in your arm, by central line in a vein, or by mouth, before your therapy begins with docetaxel plus carboplatin. Dexamethasone will help decrease bone marrow inflammation. You will also be given a colony stimulating factor (when the doctor thinks it is needed) to help maintain your white blood cell count to help decrease any chance of infection. Colony stimulating factor will be given as a subcutaneous injection (under the skin), at the discretion of the treating physician, during therapy.

You will have about 2-3 tablespoons of blood drawn at the beginning of each cycle of therapy for routine blood tests and blood tests for cancer markers. You will be asked about any medications you are currently taking.

At the end of the first 2 cycles of therapy, you will have some or all of the scans (performed during the screening visit) repeated to evaluate your disease. If your disease is responding well to the therapy, you will continue on docetaxel plus carboplatin for 2 more cycles. In this case, you will continue receive the study combination until your doctor thinks you have received the most benefit. You will then be followed with some or all of the scans (performed during the screening visit) every 2 months unless your cancer progresses (gets worse) or until you begin on a new therapy after your treatment has ended on this study.

If you are already taking hormone therapy with an luteinizing hormone-releasing hormone (LHRH) agonist (such as Lupron or Zoladex) , you will continue taking these medications. If you are taking an anti-androgen drug (such as Casodex), you should stop taking it.

If your cancer is progressing after having had a maximal response, if your disease does not respond after 2 courses of therapy, or if you are not able to tolerate some side effects of docetaxel plus carboplatin, your chemotherapy will be switched to etoposide plus cisplatin. If this is the case, etoposide plus cisplatin will be given to you by a vein in your arm or central line in a vein. You will receive this therapy combination once a day (etoposide over 60 minutes and cisplatin over 2 hours) for the first 3 days during each cycle of therapy, and then therapy will be repeated every 3 to 4 weeks.

Therapy with etoposide plus cisplatin will be continued as long as your cancer responds well to this therapy and you are not experiencing any intolerable side effects. If you experience any side effects, your dose of etoposide plus cisplatin may be decreased. This treatment combination may be given on an inpatient basis.

You will be removed from this study if your disease gets worse or you experience any intolerable side effects.

If you come off this study because you completed therapy, your disease got worse, or you experienced intolerable side effects, you will have an end-of-study visit. During this visit, you will have blood drawn (about 3 tablespoons) for routine tests. You will have a complete physical exam, including measurement of your vital signs. You will also have your complete medical history recorded and you will be asked about any medications you are currently taking. You will have imaging scans to evaluate your disease (similar to those at screening) if they have not been done in the last 28 days.

Once you are no longer on this study, the research staff will periodically check up on you (about every 6 months). This update will consist of a phone call, an e-mail, or a review of your medical and/or other records. No clinic visits or additional diagnostic studies are required by the study. If contacted by phone, the call would only last a few minutes.

This is an investigational study. Carboplatin, docetaxel, etoposide, and cisplatin are all commercially available and approved by the FDA. Up to 120 patients will take part in this multicenter study. Up to 90 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have androgen independent Stage IV prostate cancer, with anaplastic features as defined by at least one of the following: a) Histologic evidence of small cell(pure/mixed), locally advanced or metastatic; b) Any of the following at Dx: exclusive visceral mets, predominant lytic mets, bulky ( >/= 5 cm) lymphadenopathy, or bulky ( >/= 5 cm) high-grade (Gleason >/= 8) tumor mass in the prostate/pelvis c) Low prostate-specific antigen (PSA) at diagnosis (Dx) + high volume bone mets.
2. (#1 cont'd) d) Neuroendocrine markers in histology (+ Chromogranin A and/or Synaptophysin) or serum (abnl high serum Chromogranin A or Bombesin) at Dx or at progression plus any of the following: elevated serum lactate dehydrogenase (LDH), malignant HyperCa+, or elevated serum Carcinoembryonic Antigen (CEA) in the absence of other etiologies. e) Short interval (< 6 months) to androgen-independent progression following initiation of hormonal therapy with or without presence of neuroendocrine markers.
3. Patients with small cell carcinoma on histology are not required to have received prior androgen deprivation therapy (ADT). All other patients must have evidence of disease progression while on ADT or an unsatisfactory response to >/= 1 month of castration, as defined by lack of symptom control and/or serum tumor marker response of < 20% (confirmed by a second value drawn on a different day).
4. Zubrod performance status of </= 2.
5. Normal EKG or, if EKG is suggestive of cardiomyopathy, patient has a resting Left Ventricular Ejection Fraction (LEVF) >/= 50% within 4 months.
6. Patient has all of the following pretreatment laboratory data within 14 days before registration: • Absolute neutrophil count (ANC) >=1,500/mm^3.(unless due to bone marrow infiltration by tumor, in which case ANC >/= 500/mm^3 are allowed). • Platelets >=100,000/mm^3 (unless due to bone marrow infiltration by tumor, in which case platelets >/= 20,000/mm^3 are allowed)
7. (#7 cont'd) • Total bilirubin </= 2 mg/dl; if greater, conjugated bilirubin should be <= 1.0 mg/dL, • serum glutamate pyruvate transaminase (SGPT) (ALT) and/or serum glutamate oxaloacetate transaminase (SGOT) (AST) </= 4 times the upper limit of normal (ULN). • Creatinine clearance >/= 40 (either measured or calculated by Cockcroft formula) • Castrate levels of serum testosterone (</= 50ng/mL) if no small cell elements on histology. (If small cell, testosterone > 50ng/mL)
8. Patient has given voluntary written informed consent before performance of any study-related procedure not part of standard medical care.

Exclusion Criteria:

1. Immunotherapy or chemotherapy within four weeks (nitrosoureas within six weeks) of registration.
2. 2 or more prior chemotherapy regimens (ketoconazole, aminoglutethimide or dutasteride do not count as chemotherapy for this trial).
3. Prior Platinum, Etoposide, or Taxane-based therapy that was completed less than 6 months from registration.
4. Samarium-153 within four weeks of registration, or Strontium-89 within 12 weeks of registration. Patients who have received 2 or more doses of bone-seeking radioisotopes are not eligible.
5. Patient has not recovered from all serious toxic effects of previous chemotherapy, radiation or antibody therapy, or from previous major surgery.
6. Patients with symptomatic and untreated brain metastases or central nervous system disease will be excluded. Patients with untreated, asymptomatic brain metastasis (not requiring corticosteroid treatment for control of central nervous system (CNS) symptoms) may be eligible, at the discretion of the MDACC Principal Investigator. Patients with treated brain metastases are eligible.
7. Patient with significant atherosclerotic disease, as defined by: a) myocardial infarction within six months of enrollment. Current uncontrolled/unstable angina pectoris or electrocardiographic evidence of acute ischemia b) clinically significant ventricular arrhythmias c) symptomatic congestive heart failure (NYHA Class III)
8. Patient has >= Grade 2 peripheral neuropathy.
9. Patient has renal insufficiency with cranial cruciate ligament (CrCL) < 40 ml/min with non-correctable etiologies.
10. Patient has an uncontrolled intercurrent illness (e.g., active infection).
11. Patient has another serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the patient's ability to provide informed consent or with the completion of treatment according to this protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Aparicio, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of California-San Francisco, San Francisco, California
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Aparicio AM, Harzstark AL, Corn PG, Wen S, Araujo JC, Tu SM, Pagliaro LC, Kim J, Millikan RE, Ryan C, Tannir NM, Zurita AJ, Mathew P, Arap W, Troncoso P, Thall PF, Logothetis CJ. Platinum-based chemotherapy for variant castrate-resistant prostate cancer. Clin Cancer Res. 2013 Jul 1;19(13):3621-30. doi: 10.1158/1078-0432.CCR-12-3791. Epub 2013 May 6. PMID 23649003
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled between June 2006 and October 2010 at The University of Texas (UT) MD Anderson Cancer Center (MDACC).
Pre-assignment Details: Of the 121 participants enrolled, seven were ineligible and excluded. Another participant was eligible but withdrew before treatment.
Groups:
- Chemotherapy First-Line Chemo (CD) + Second-Line (EP): First-Line (CD) Chemotherapy: Carboplatin area under the curve (AUC) = 5, intravenous (IV) over 30 minutes and Docetaxel 75 mg/m^2 IV over 60 minutes, Day 1. Repeated every 3 weeks. Colony stimulating factors given prophylactically per National Comprehensive Cancer Network (NCCN) guidelines.
  Second-Line (EP) Chemotherapy: Etoposide 120 mg/m^2 daily for 3 days and Cisplatin 25 mg/m^2 for 3 days with adequate intravenous hydration mannitol diuresis and supportive care (antiemetics). Repeated every 3 weeks.
Period: First-Line Chemo
Arm/Group | Chemotherapy First-Line Chemo (CD) + Second-Line (EP)
Started | 113
Completed | 105
Not Completed | 8
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 7
Period: Second-Line
Arm/Group | Chemotherapy First-Line Chemo (CD) + Second-Line (EP)
Started | 105
Completed | 74
Not Completed | 31
Not completed — Physician/Patient Decision | 31

BASELINE CHARACTERISTICS:
Population: Eligibile population treated.
Groups:
- First-Line CD + Second-Line EP: First-Line (CD) Chemotherapy: Carboplatin area under the curve (AUC) = 5, intravenous (IV) over 30 minutes and Docetaxel 75 mg/m^2 IV over 60 minutes, Day 1. Repeated every 3 weeks. Colony stimulating factors given prophylactically per National Comprehensive Cancer Network (NCCN) guidelines.
  Second-Line (EP) Chemotherapy: Etoposide 120 mg/m^2 daily for 3 days and Cisplatin 25 mg/m^2 for 3 days with adequate intravenous hydration mannitol diuresis and supportive care (antiemetics). Repeated every 3 weeks.
Arm/Group | First-Line CD + Second-Line EP
Number analyzed (Participants) | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 50
Age, Continuous [Median (Full Range); unit: years] | 64 [39 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 113
Region of Enrollment [Number; unit: participants]
  United States | 113

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression (TTP)
Description: TTP defined as time of registration on study till disease progression. Disease status evaluated at the end of course 1 (up to 84 days after day 1 of cycle 1) and at the end of course 2 (up to 168 days after day 1 of cycle 1).
Time Frame: Baseline to evaluation at end of course 2 (up to 168 days) then every 2 months for disease progression. Follow up every 6 months and overall study period was six and half years.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- First-Line: Carboplatin + Docetaxel: Carboplatin area under the curve (AUC) = 5, intravenous (IV) over 30 minutes and Docetaxel 75 mg/m^2 IV over 60 minutes, Day 1 repeated every 3 weeks.
- Second-Line: Etoposide + Cisplatin: Etoposide 120 mg/m^2 daily for 3 days and Cisplatin 25 mg/m^2 for 3 days with adequate intravenous hydration mannitol diuresis and supportive care (antiemetics). Repeated every 3 weeks.
Arm/Group | First-Line: Carboplatin + Docetaxel | Second-Line: Etoposide + Cisplatin
Number analyzed (Participants) | 113 | 74
months | 5.1 [4.2 to 6.0] | 3.0 [1.6 to 3.5]
Statistical Analysis 1: Comparison: First-Line: Carboplatin + Docetaxel vs Second-Line: Etoposide + Cisplatin; Disease status evaluated at the end of course 1 & the end of course 2. Primary outcomes are response, defined as the absence of disease progression, and the time to a serious adverse event (SAE), defined as grade 3 or 4 neurotoxicity or death. Bayesian probability model & decision rules used to monitor patient outcomes; Test type: Superiority or Other; p < 0.005, Bayesian probability model — Stoppage of trial early if 1) probability of response with the frontline treatment DC in the 1st 2 courses is unacceptably low compared to a target of 30% Pr(p1*p2 > .30|data) < 0.005, or 2) risk of a SAE is unacceptably high Pr(m > m* |data) < 0.001; Operating Characteristics of futility monitoring rule 1 & safety monitoring rule 2 applied simultaneously for frontline treatment DC in courses 1 & 2

2. Primary Outcome: Response Rate of Salvage Chemotherapy With Etoposide Plus Cisplatin Following Treatment With Docetaxel Plus Carboplatin.
Description: Response rate is the number of participants with response compared to total. Response defined as the absence of disease progression compared to the participant's baseline evaluation, and the time to a serious adverse event (SAE), defined as grade 3 or 4 neurotoxicity or death.
Time Frame: Evaluated at the end of course 1 (up to 84 days after day 1 of cycle 1) and at the end of course 2 (up to 168 days after day 1 of cycle 1)
Population: 74 of the 105 participants received second-line EP on study; the remainder withdrew from the study at their physician's or their own request. 2 participants died after course 1 of EP.
Measure: Number; unit: participants
Groups:
- Second-Line: EP, Course 1; Second-Line: EP, Course 2: Etoposide 120 mg/m^2 daily for 3 days and Cisplatin 25 mg/m^2 for 3 days with adequate intravenous hydration mannitol diuresis and supportive care (antiemetics). Repeated every 3 weeks.
Arm/Group | Second-Line: EP, Course 1 | Second-Line: EP, Course 2
Number analyzed (Participants) | 74 | 41
participants | 43 | 24

ADVERSE EVENTS:
Time Frame: One therapy course consists of two (2) cycles, each cycle is defined as 21 days. Safety stopping rule assessed at the end of one course Docetaxel + Carboplatin and at the end of one course Etoposide + Cisplatin. Toxicity data collected for all cycles.
Groups:
- First-Line: Carboplatin + Docetaxel: Carboplatin area under the curve (AUC) = 5, intravenous (IV) over 30 minutes and Docetaxel 75 mg/m2 IV over 60 minutes, Day 1 repeated every 3 weeks
- Second Line: Etoposide + Cisplatin: Etoposide 120 mg/m2 daily for 3 days and Cisplatin 25 mg/m2 for 3 days with adequate intravenous hydration mannitol diuresis and supportive care (antiemetics), Repeated every 3 weeks.
Arm/Group | First-Line: Carboplatin + Docetaxel | Second Line: Etoposide + Cisplatin
All-Cause Mortality (participants affected / at risk) | 3/113 | 1/74
Serious Adverse Events (participants affected / at risk) | 18/113 | 10/74
Other Adverse Events (participants affected / at risk) | 112/113 | 58/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First-Line: Carboplatin + Docetaxel (N=113) | Second Line: Etoposide + Cisplatin (N=74)
Hyperbilirubin (Metabolism and nutrition disorders) | 1 (1) | 0
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0
Disseminated Intravascular Coagulation (Vascular disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0
Edema: Limb (Blood and lymphatic system disorders) | 1 (1) | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Lung pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Upper airway infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Rigors/chills (General disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Thrombosis/embolism (Vascular disorders) | 1 (1) | 2 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Vasovagal episode (Cardiac disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First-Line: Carboplatin + Docetaxel (N=113) | Second Line: Etoposide + Cisplatin (N=74)
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 62 (129) | 22 (36) — Grade 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 27 (45) | 17 (27)
ALT elevated (Metabolism and nutrition disorders) | 15 (25) | 2 (3)
Anorexia (Gastrointestinal disorders) | 8 (15) | 4 (4)
AST elevated (Metabolism and nutrition disorders) | 28 (42) | 10 (10)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 9 (15) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (36) | 15 (30)
Constipation (Gastrointestinal disorders) | 13 (15) | 4 (4)
Creatinine (Metabolism and nutrition disorders) | 12 (17) | 13 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 42 (68) | 21 (24)
Edema (Blood and lymphatic system disorders) | 18 (34) | 12 (12) — Head and neck, limbs, trunk/genital, viscera
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 99 (359) | 44 (125)
Fever (General disorders) | 11 (13) | 3 (3)
Hair Loss/Alopecia (Skin and subcutaneous tissue disorders) | 15 (16) | 0 (0)
Hemoglobin (Metabolism and nutrition disorders) | 76 (211) | 47 (139)
Infection with normal ANC (Infections and infestations) | 7 (8) | 3 (4)
Injection Site Reaction/Extravasation Changes (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (1)
Leukocytes (Total WBC) (Blood and lymphatic system disorders) | 70 (204) | 27 (60)
Hypomagnesemia (Metabolism and nutrition disorders) | 38 (67) | 35 (66)
Nail Changes (Skin and subcutaneous tissue disorders) | 18 (20) | 1 (1)
Nausea (Gastrointestinal disorders) | 75 (216) | 34 (64)
Neuropathy: Sensory (Nervous system disorders) | 45 (79) | 16 (23)
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 62 (129) | 22 (96)
Pain (General disorders) | 17 (23) | 5 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (11) | 5 (8)
Platelets (Blood and lymphatic system disorders) | 53 (124) | 42 (124)
Hyperkalemia (Metabolism and nutrition disorders) | 21 (30) | 9 (13)
Hyponatremia (Metabolism and nutrition disorders) | 26 (45) | 25 (42)
Dysgeusia (Gastrointestinal disorders) | 6 (14) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Vomitting (Gastrointestinal disorders) | 33 (97) | 13 (24)
Watery Eye (Eye disorders) | 26 (45) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 56 (139) | 29 (31)
Mucositis (Gastrointestinal disorders) | 17 (34) | 9 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No